CLINICAL TRIAL: NCT04868916
Title: Prospective Observational Study to Estimate the Genotype and Phenotype of Japanese Patients With X-linked Retinitis Pigmentosa Associated With Pathogenic Variants in Retinitis Pigmentosa GTPase Regulator (RPGR)
Brief Title: An Observational Study of Japanese Participants With X-linked Retinitis Pigmentosa
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108926; 74765340RPG0001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: X-Linked Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with X-Linked Retinitis Pigmentosa (XLRP): Participants with confirmed diagnosis of XLRP associated with pathogenic variants in retinitis pigmentosa GTPase regulator (RPGR) in the Japanese population will be enrolled in the study and the data will be collected and observed. The primary data source for this study will be the medical records of each participant.

SUMMARY:
The purpose of the study is to identify a cohort of Japanese participants with X-linked retinitis pigmentosa (XLRP) associated with pathogenic variants in the retinitis pigmentosa GTPase regulator (RPGR) gene and to investigate their associated phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Have RPGR-associated retinal dystrophy
* Are able to give informed consent or assent, with the guidance of their parent/guardian where appropriate
* Are able to undertake age-appropriate clinical assessments as specified in the protocol

Exclusion Criteria:

* Are unable or unwilling to undertake consent or clinical testing
* Participated in another research study and had intraocular surgery within 3 months of screening
* Significant ophthalmologic diseases

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population consists of Japanese participants with X-linked retinitis pigmentosa (XLRP) associated with pathogenic variants in retinitis pigmentosa GTPase regulator (RPGR).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Visual Function | Up to Day 30
  Visual function will be assessed using visual acuity.
Retinal Structure | Up to Day 30
  Retinal structure will be assessed using spectral domain optical coherence tomography (SDOCT).
Retinal Function | Up to Day 30
  Retinal function will be assessed using static visual field testing.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- National Hospital Organization Tokyo Medical Center, Tokyo, Japan

REFERENCES:
- [Derived] Fujinami-Yokokawa Y, Yang L, Joo K, Tsunoda K, Liu X, Kondo M, Ahn SJ, Li H, Park KH, Tachimori H, Miyata H, Woo SJ, Sui R, Fujinami K. Occult Macular Dysfunction Syndrome: Identification of Multiple Pathologies in a Clinical Spectrum of Macular Dysfunction with Normal Fundus in East Asian Patients: EAOMD Report No. 5. Genes (Basel). 2023 Sep 26;14(10):1869. doi: 10.3390/genes14101869. PMID 37895218